CLINICAL TRIAL: NCT01583725
Title: Functional Brain Imaging and Appetite-Related Hormones Pre and Post Obesity Surgery
Brief Title: fMRI and Appetite-Related Hormones Pre and Post Obesity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Obesity and Nutrition Research Center (Other)
Collaborators: Columbia University (Other); St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Principal Investigator, Dr. Allan Geliebter, Principal Investigator, New York Obesity and Nutrition Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-101
Record Dates: First submitted 2012-03-09; First posted 2012-04-24 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Weight loss; fMRI; gut peptides
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Roux-en-Y Gastric Bypass (Experimental): 30 subjects who plan to undergo Roux-en-Y Gastric Bypass bariatric surgery. Liquid meal responses and Behavioral fMRI responses to food-cues will be assessed before surgery (T1), 3 months (T2) and 18 months (T3) after surgery.
  Interventions: Procedure: Liquid meal responses; Behavioral: fMRI responses to food-cues
- Gastric Banding (Lap-band) (Experimental): 30 subjects who plan to undergo Gastric Banding bariatric surgery. Liquid meal responses and Behavioral fMRI responses to food-cues will be assessed before surgery (T1), 3 months (T2) and 18 months (T3) after surgery.
  Interventions: Procedure: Liquid meal responses; Behavioral: fMRI responses to food-cues
- Formula Diet Weight Loss (Experimental): 30 subjects who plan to begin a formula diet to lose weight. Liquid meal responses and Behavioral fMRI responses to food-cues will be assessed before subjects undertake a 12-week weight loss intervention (T1), at the end of the weight loss intervention (T2) and 18 months after they completed the weight loss intervention(T3).
  Interventions: Procedure: Liquid meal responses; Behavioral: fMRI responses to food-cues
- No Treatment (Experimental): 30 subjects who do not undergo any treatment for weight loss. Liquid meal responses and Behavioral fMRI responses to food-cues will be assessed at baseline (T1) and at 3 months (T2) and 18 months (T3) later.
  Interventions: Procedure: Liquid meal responses; Behavioral: fMRI responses to food-cues
- Sleeve Gastrectomy Surgery (Experimental): 30 subjects who plan to undergo Sleeve Gastrectomy bariatric surgery. Liquid meal responses and Behavioral fMRI responses to food-cues will be assessed before surgery (T1), 3 months (T2) and 18 months (T3) after surgery.
  Interventions: Procedure: Liquid meal responses; Behavioral: fMRI responses to food-cues

INTERVENTIONS:
Procedure: Liquid meal responses — Subject ingests a meal-replacement shake and gut peptide levels are measured before and after intake.
  Other Names: Meal replacement shake is the product Glytrol.
Behavioral: fMRI responses to food-cues — Subjects undergo a 40 min fMRI neuroimaging session while receiving auditory and visual food cues.
  Other Names: Food cue responses

SUMMARY:
The investigators are looking at the differences in appetite and obesity between weight loss participants and patients undergoing bariatric surgery.

Obese persons between the ages of 18 & 65 are eligible to participate in this study, whether or not they intend to undergo bariatric surgery.

DETAILED DESCRIPTION:
Currently, the only effective long term treatment for severe obesity is bariatric surgery.2 Nearly 200,000 procedures are performed each year, with this number increasing rapidly.3 However, the mechanisms of reduced food intake and weight loss after obesity surgery, particularly Rouen-Y gastric bypass (RYGB), are not well understood. This study utilizes functional magnetic resonance imaging (fMRI) and measures of appetite-related gut peptide levels pre and post bariatric surgery to investigate the neurological and hormonal mechanisms involved in initiation and termination of meals.

The general objective is to better understand the physiological changes resulting in weight loss from obesity surgery, particularly Roux-en-Y gastric bypass (RYGB). The main hypothesis is that the differential mechanisms of action in RYGB will alter the signals involved in the initiation and termination of meals, reflected by changes in both peptide hormone levels and regional brain activity in response to foods. The investigators anticipate that the trigger for meal initiation by potent food stimuli will be diminished following RYGB, as indicated by reduced brain activation in areas associated with food reward and motor planning, including the orbitofrontal cortex (OFC). RYGB will be compared to: a. Gastric Banding (GB), representing the restrictive component of surgery, which itself enhances fullness, but in the absence of any rerouting of the gut, should result in fewer changes in gut peptide levels and brain activation; b. Weight Loss (WL) on a formula diet over 3 mo, which represents the weight loss component of surgery; and c. No Treatment (NT), a general control, with no gastric restriction or weight loss. These group comparisons will help parse the contributions of RYGB surgery to weight loss.

The plan is to study clinically severe obese subjects (S's) pre surgery, and at 3 and 18 mo post surgery. The investigators will examine: 1) fMRI brain activation in response to food stimuli and 2) appetite-related gut peptide levels before and following a fixed meal prior to the fMRI. The findings should reveal potential mechanisms associated with the changes in appetite, eating behaviors, and body weight, both during the rapid weight loss phase at 3 mo post surgery as well as when weight typically stabilizes at a nadir at 18 mo post surgery. The investigators plan to enroll 160 patients: 40 with RYGB, 40 GB, 40 WL, and 40 NT (4-arm study). S's will be within the BMI range of 40-50 and matched across groups for BMI, gender (3:1, f:m), and BED status.

ELIGIBILITY:
Inclusion Criteria:

* BMI range 35-50 kg/m^2

Exclusion Criteria:

* diabetes,
* smoking,
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in brain activation in response to visual and auditory food cues | 3 mo pre-surgery and 3 and 18 mo post-surgery
  Measures of brain brain activation in areas associated with food reward and motor planning, including the orbitofrontal cortex (OFC). Over the course of 40-min fMRI scans, we will compare change in activation from 3 mo pre-surgery to 3 and 18 mo post-surgery, and predict a post-surgical decrease in activation in such regions.

SECONDARY OUTCOMES:
Anthropometrics and Body Composition | 3 mo pre-surgery and 3 and 18 mo post-surgery
  Height and weight will be assessed using a stadiometer and digital scale. Sagittal diameter and waist and hip circumferences, as well as maximum supine width, will be measured. Waist circumference will be measured. Air displacement (Bioelectrical impedance analyses) will also be performed to obtain lean and fat mass. Weights, BMI, and body composition will confirm that the four obese groups are similar at baseline and provide estimates of changes in body fat following treatment.
Mood Measures | 3 mo pre-surgery and 3 and 18 mo post-surgery
  We will administer relevant psychological instruments to assess Mood:
  The Inventory of Depressive Symptomatology-Self Report (IDS-SR)will be assessed at 3mo pre-surgery, 3mo, 6mo and 18mo post surgery.
Change in appetite-related gut peptide levels | 3 mo pre-surgery and 3 and 18 mo post-surgery
  We will measure changes in appetite-related gut peptide levels before and following a fixed meal prior to the fMRI. This will be assessed via blood plasma samples taken on 3 occasions: 3 mo pre-surgery, 3 mo post-surgery, and 18 mo post-surgery. At each session, there will be multiple time points: -15, 0, 15, 30, 60, and 90 minutes before/after ingestion of a meal replacement shake.
Eating Behavior | 3 mo pre-surgery and 3 and 18 mo post-surgery
  We will administer relevant psychological instruments to assess Eating Behavior:including Eating Disorder Examination (EDE) to diagnose BED; Binge Eating Scale (BES), correlated with BED status; eating-related behavior (DEBQ - Restraint, Emotional, and Externality subscales); and dietary intake (24-Hour Food Recall).

CONTACTS AND LOCATIONS:
Overall Officials: Allan Geliebter, PhD, Principal Investigator — New York Obesity Nutrition Research Center, St. Luke's-Roosevelt Hospital, Columbia University
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Background] Ongur D, Price JL. The organization of networks within the orbital and medial prefrontal cortex of rats, monkeys and humans. Cereb Cortex. 2000 Mar;10(3):206-19. doi: 10.1093/cercor/10.3.206. PMID 10731217
- [Background] Le DS, Pannacciulli N, Chen K, Del Parigi A, Salbe AD, Reiman EM, Krakoff J. Less activation of the left dorsolateral prefrontal cortex in response to a meal: a feature of obesity. Am J Clin Nutr. 2006 Oct;84(4):725-31. doi: 10.1093/ajcn/84.4.725. PMID 17023697
- [Background] Le DS, Pannacciulli N, Chen K, Salbe AD, Del Parigi A, Hill JO, Wing RR, Reiman EM, Krakoff J. Less activation in the left dorsolateral prefrontal cortex in the reanalysis of the response to a meal in obese than in lean women and its association with successful weight loss. Am J Clin Nutr. 2007 Sep;86(3):573-9. doi: 10.1093/ajcn/86.3.573. PMID 17823419
- [Background] Rosenbaum M, Leibel RL, Hirsch J. Obesity. N Engl J Med. 1997 Aug 7;337(6):396-407. doi: 10.1056/NEJM199708073370606. No abstract available. PMID 9241130
- [Background] Whitson BA, Leslie DB, Kellogg TA, Maddaus MA, Buchwald H, Billington CJ, Ikramuddin S. Entero-endocrine changes after gastric bypass in diabetic and nondiabetic patients: a preliminary study. J Surg Res. 2007 Jul;141(1):31-9. doi: 10.1016/j.jss.2007.02.022. PMID 17574036
- [Background] Korner J, Bessler M, Cirilo LJ, Conwell IM, Daud A, Restuccia NL, Wardlaw SL. Effects of Roux-en-Y gastric bypass surgery on fasting and postprandial concentrations of plasma ghrelin, peptide YY, and insulin. J Clin Endocrinol Metab. 2005 Jan;90(1):359-65. doi: 10.1210/jc.2004-1076. Epub 2004 Oct 13. PMID 15483088
- [Background] le Roux CW, Welbourn R, Werling M, Osborne A, Kokkinos A, Laurenius A, Lonroth H, Fandriks L, Ghatei MA, Bloom SR, Olbers T. Gut hormones as mediators of appetite and weight loss after Roux-en-Y gastric bypass. Ann Surg. 2007 Nov;246(5):780-5. doi: 10.1097/SLA.0b013e3180caa3e3. PMID 17968169
- [Background] Sorbara M, Geliebter A. Body image disturbance in obese outpatients before and after weight loss in relation to race, gender, binge eating, and age of onset of obesity. Int J Eat Disord. 2002 May;31(4):416-23. doi: 10.1002/eat.10046. PMID 11948646
- [Background] Jirik-Babb P, Geliebter A. Comparison of psychological characteristics of binging and nonbinging obese, adult, female outpatients. Eat Weight Disord. 2003 Jun;8(2):173-7. doi: 10.1007/BF03325009. PMID 12880197
- [Background] Erdmann J, Topsch R, Lippl F, Gussmann P, Schusdziarra V. Postprandial response of plasma ghrelin levels to various test meals in relation to food intake, plasma insulin, and glucose. J Clin Endocrinol Metab. 2004 Jun;89(6):3048-54. doi: 10.1210/jc.2003-031610. PMID 15181097
- [Background] Marzullo P, Verti B, Savia G, Walker GE, Guzzaloni G, Tagliaferri M, Di Blasio A, Liuzzi A. The relationship between active ghrelin levels and human obesity involves alterations in resting energy expenditure. J Clin Endocrinol Metab. 2004 Feb;89(2):936-9. doi: 10.1210/jc.2003-031328. PMID 14764817
- [Background] Hosoda H, Doi K, Nagaya N, Okumura H, Nakagawa E, Enomoto M, Ono F, Kangawa K. Optimum collection and storage conditions for ghrelin measurements: octanoyl modification of ghrelin is rapidly hydrolyzed to desacyl ghrelin in blood samples. Clin Chem. 2004 Jun;50(6):1077-80. doi: 10.1373/clinchem.2003.025841. No abstract available. PMID 15161728
- [Background] Liu J, Prudom CE, Nass R, Pezzoli SS, Oliveri MC, Johnson ML, Veldhuis P, Gordon DA, Howard AD, Witcher DR, Geysen HM, Gaylinn BD, Thorner MO. Novel ghrelin assays provide evidence for independent regulation of ghrelin acylation and secretion in healthy young men. J Clin Endocrinol Metab. 2008 May;93(5):1980-7. doi: 10.1210/jc.2007-2235. Epub 2008 Mar 18. PMID 18349056
- [Background] Geliebter A, Ladell T, Logan M, Schneider T, Sharafi M, Hirsch J. Responsivity to food stimuli in obese and lean binge eaters using functional MRI. Appetite. 2006 Jan;46(1):31-5. doi: 10.1016/j.appet.2005.09.002. Epub 2005 Dec 20. PMID 16364498
- See also: New York Obesity Nutrition Research Center website — http://www.nyorc.org/